CLINICAL TRIAL: NCT06997913
Title: Adjuvant Immunotherapy Combined With ChemoRadiation for Patients With High-risk Resectable Extrahepatic Cholangiocarcinoma（AICRC）
Acronym: AICRC
Status: Enrolling by invitation | Type: Observational
Sponsor: Hengchao Yu (Other)
Responsible Party: Sponsor-Investigator, Hengchao Yu, Professor, The First Affiliated Hospital of Air Force Medicial University
Organization: The First Affiliated Hospital of Air Force Medicial University (Other)
Other Study IDs: KY20242343-F-1
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Lymph Node Metastasis; Neurovascular Invasion; Pathology Showed R1 Resection
Keywords: extrahepatic cholangiocarcinoma; high-risk recurrence populations; adjuvant chemoradiotherapy combined with immunotherapy
MeSH Terms: conditions — Lymphatic Metastasis; Cholangiocarcinoma | interventions — Chemoradiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — tumor tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adjuvant chemoradiotherapy combined with immunotherapy: This is a single-arm, prospective clinical study designed to evaluate the efficacy and safety of tislelizumab injection combined with capecitabine and radiotherapy as first-line adjuvant therapy for high-risk recurrence populations after extrahepatic cholangiocarcinoma (ECC) resection.
  Interventions: Combination Product: Adjuvant Immunotherapy Combined With ChemoRadiation for Patients With High-risk resectable Extrahepatic Cholangiocarcinoma（AICRC）

INTERVENTIONS:
Combination Product: Adjuvant Immunotherapy Combined With ChemoRadiation for Patients With High-risk resectable Extrahepatic Cholangiocarcinoma（AICRC） — The purpose of this prospective, observational study is to investigate whether adjuvant chemoradiotherapy combined with immunotherapy for high-risk recurrence populations after extrahepatic cholangiocarcinoma resection can improve patients' recurrence-free survival. The primary study endpoint of this prospective study is the 2-year recurrence-free survival.

SUMMARY:
The purpose of this prospective, observational study is to investigate whether adjuvant chemoradiotherapy combined with immunotherapy for high-risk recurrence populations after extrahepatic cholangiocarcinoma resection can improve patients' recurrence-free survival. The primary study endpoint of this prospective study is the 2-year recurrence-free survival.

DETAILED DESCRIPTION:
This is a single-arm, prospective clinical study designed to evaluate the efficacy and safety of tislelizumab injection combined with capecitabine and radiotherapy as first-line adjuvant therapy for high-risk recurrence populations after extrahepatic cholangiocarcinoma (ECC) resection. The study will enroll patients with ECC who have not received prior systemic therapy. The primary endpoint is the 2-year recurrence-free survival rate (2y-RFS), with a planned enrollment of approximately 65 subjects.

After providing full informed consent, eligible patients will receive treatment with tislelizumab injection combined with capecitabine and radiotherapy. Each study treatment cycle is 3 weeks, and treatment will continue until the criteria for terminating study treatment are met.

Treatment regimen for the treatment group:

1. Tislelizumab injection: 200 mg via intravenous infusion (D1), administered every 21 days (Q3W), with maintenance treatment for at least half a year or until disease progression.
2. Capecitabine: 1000 mg/m², twice daily (D1-14), administered every 21 days (Q3W) for a total of 6 treatment cycles.
3. Radiotherapy: 50Gy to regional lymph nodes and preoperative tumor bed.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70 years;
2. Primary resectable extrahepatic cholangiocarcinoma proved by pathology which underwent radical surgery;
3. Pathology indicates R0 with N1 or Neurovascular invasion; or R1;
4. ECOG PS 0-1;
5. Adequate hematologic, hepatic and renal function: ANC ≥ 1.5x10^9/L, Hb ≥ 80g/L, PLT ≥ 100 x10^9/L, albumin ≥ 28g/L, total bilirubin < 1.5×ULN, ALT and AST < 2.5×ULN, CREA<1.5×ULN;
6. No anti-tumor treatment before radical resection, including radiotherapy and chemotherapy, targeted therapy and immunotherapy；
7. At least 6 months of life expectancy.

Exclusion Criteria:

1. Diagnosis of other malignant diseases outside the biliary tract within 5 years before the first administration (excluding radically cured skin basal cell carcinoma, skin squamous cell carcinoma, and/or radically excised carcinoma in situ);
2. Pregnant or breastfeeding women, or expecting to conceive or father children within the projected duration of the trial;
3. With purulent, infected or delayed healed wounds;
4. Have thromboembolism in the past 6 months, including myocardial infarction, unstable angina, stroke or transient ischemic attack, pulmonary embolism, deep vein thrombosis;
5. An active autoimmune disease that requires systemic treatment (such as the use of disease-relieving drugs, glucocorticoids, or immunosuppressive agents) occurred within 2 years before the first administration. Alternative therapies (such as thyroxine, insulin, or physiological glucocorticoids for adrenal or pituitary insufficiency) are not considered systemic treatments. Known history of primary immunodeficiency. Only patients with positive autoimmune antibodies need to confirm whether there are autoimmune diseases based on the judgment of the investigator;
6. Are receiving systemic glucocorticoid therapy (excluding nasal spray, inhaled or other local glucocorticoids) or any other form of immunosuppressive therapy within 4 weeks before the first administration of the study. Note: Physiological doses of glucocorticoids are allowed (≤10 mg/day prednisone or equivalent drugs);
7. Have other uncontrollable comorbidities;
8. Infection of HIV, known syphilis requiring treatment;
9. Uncontrollable hypertension, systolic pressure>140mmHg or diastolic pressure>90mmHg after best medical care, or history of hypertensive crisis or hypertensive encephalopathy;
10. Symptomatic congestive heart failure (NYHA class II-IV). Symptomatic or badly-controlled arrhythmia. Congenital long QT syndrome or modified QTc>500ms upon screening;
11. Have active autoimmune diseases that require systemic treatment within 2 years before enrolment;
12. Active tuberculosis, having antituberculosis therapy at present or within 1 year;
13. The medical history or disease evidence, abnormal treatment or laboratory test values that may interfere with the test results, prevent the subject from participating in the study, or the investigator believes that it is not suitable for inclusion in the group. The investigator believes that there are other potential risks and is not suitable for participation；

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients With High-risk resectable Extrahepatic Cholangiocarcinoma
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
2-year recurrence-free survival rate | 2 Year
  The target population is enrolled and receives postoperative adjuvant therapy according to the study protocol, the recurrence-free survival status of patients will be observed at 2 years.

SECONDARY OUTCOMES:
2-year overall survival rate | 2 Year
  The target population is enrolled and receives postoperative adjuvant therapy according to the study protocol, the overall survival status of patients will be observed at 2 years.
Incidence of adverse events | 2 Year
Completion rate of treatment | 2 Year

CONTACTS AND LOCATIONS:
Overall Officials: Lin Wang Professor.Wang, Doctor of Medicine(M.D.), Study Chair — Department of Hepatobiliary Surgery, the First Affiliated Hospital of Air Force Military Medical University
Locations (1):
- Department of Hepatobiliary Surgery, the First Affiliated Hospital of Air Force Military Medical University, XiAn, Shanxi, China

IPD SHARING:
Plan to Share IPD: Yes
The survival data of the Patients With High-risk resectable Extrahepatic Cholangiocarcinoma after treatment
Supporting Information: Study Protocol
Time Frame: 2 Year
Access Criteria: All medical workers